CLINICAL TRIAL: NCT04208191
Title: Strengthening People-centered Accessibility, Respect, and Quality for Maternal Health and Family Planning Services in Nairobi, Kenya
Brief Title: Quality Improvement Project for Maternal Health and Family Planning Services in Kenya
Acronym: SPARQ_QIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-18008_KenyaQI
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Maternal Health; Family Planning; Delivery
Keywords: Maternal Health; Family Planning; Quality Improvement; Person Centered Care; Kenya; Delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control - Women (No Intervention): Participants who delivered or received family planning services at a facility that was not implementing a QI project on PCC
- Intervention - Women (Experimental): Participants who delivered or received family planning services at a facility that was implementing a QI project on PCC
  Interventions: Behavioral: Quality Improvement Collaborative
- Control - Provider (No Intervention): Provider working in a facility that is not implementing a QI project on PCC
- Intervention - Provider (Experimental): Provider working in a facility that is implementing a QI project on PCC
  Interventions: Behavioral: Quality Improvement Collaborative

INTERVENTIONS:
Behavioral: Quality Improvement Collaborative — Facilities that participated in a QI collaborative to improve PCC for MH and FP services
  Arms: Intervention - Provider; Intervention - Women

SUMMARY:
Evaluation of a quality improvement (QI) collaborative aimed at improving person-centered care (PCC) for maternal health (MH) and family planning (FP) services

DETAILED DESCRIPTION:
Evaluation of a quality improvement (QI) collaborative in public facilities in Nairobi and Kiambu Counties in Kenya aimed at improving person-centered care (PCC) for maternal health (MH) and family planning (FP) services.

ELIGIBILITY:
Inclusion Criteria for Women:

* Women aged 15-49 years old
* Agreed/consented to participate
* Delivered at the facility within the last 7 days OR adopted a family planning method at their visit on day of survey
* Has a working mobile phone and specified service provider (airtel/safaricom)

Exclusion Criteria for Women:

* Not a women aged 15-49 years old
* Did no agreed/consented to participate
* Did not deliver at the facility within the last 7 days OR adopted a family planning method at their visit on day of survey
* Does not have a working mobile phone or specified service provider (airtel/safaricom)

Inclusion Criteria for Providers:

* Agreed/consented to participate
* Staff at facility

Exclusion Criteria for Providers

* Did no agreed/consent to participate
* Not staff at facility

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3354 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Person Centered Maternal Health Scale Score | Baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 2-weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 4-weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 6-weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 10-weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 24 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 26 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 30 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | About 30.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | about 31 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 31.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 32 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Maternal Health Scale Score | 32.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-100; higher the score the better the experience of care
Person Centered Family Planning Scale Score | Baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 4 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 6 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 8 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | 10 weeks post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 24 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 26 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 30 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 31 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 31.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 32 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Person Centered Family Planning Scale Score | About 32.5 months post baseline
  Survey conducted with women: self report of experiences of care. Possible range 0-43; higher the score the better the experience of care
Attitudes toward Person-Centered Care | Baseline
  Survey and In-depth interviews conducted with providers; perceptions of person-centered care
Attitudes toward Person-Centered Care | About 24 months post baseline
  Survey conducted with providers; perceptions of person-centered care
Attitudes toward Person-Centered Care | About 26 months post baseline
  Survey conducted with providers; perceptions of person-centered care
Attitudes toward Person-Centered Care | About 30 months post baseline
  Survey and In-depth interviews conducted with providers; perceptions of person-centered care
The Model for Understanding Success in Quality Survey | About 30 months post baseline
  Survey conducted with intervention providers on facility readiness to implement QI; Possible range 0-154; higher the score the more ready facility is to participate in QI activities

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Montagu, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Innovations for Poverty Action, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No